CLINICAL TRIAL: NCT03693092
Title: LAmbre™ Left Atrial Appendage Closure System Post-Market 2-5 Years Follow-Up Study
Brief Title: LAmbre™ Left Atrial Appendage Closure System Follow-Up Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LAA 2-5ys FU
Record Dates: First submitted 2018-09-30; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to conduct a continuous telephone follow-up study on subjects who had completed the one-year follow-up of the LAmbre™ left atrial appendage (LAA) system registration trial. The follow-up time was 2 years, 3 years, 4 years and 5 years after left atrial appendage closure operation, to evaluate the long-term safety and effectiveness of LAmbre™ LAA Closure System.

DETAILED DESCRIPTION:
All subjects who completed 1-year follow-up of the LAmbreTM LAA system registration trial will be conducted 2 years, 3 years, 4 years and 5 years follow-up by the telephone call.

During the follow-up, the investigator or his/her designee will use a standardized form to record the occurrence of the subject's safety events and validity endpoint by telephone，and complete the safety and efficacy summary report. The endpoints of the study included compound events, MACCE events, stroke, haemorrhage and other events.

ELIGIBILITY:
Inclusion Criteria:

- Patients who participated in the LAmbreTM Safety and Efficacy Study and completed the 1-year follow-up.

The inclusion criteria of LAmbreTM Safety and Efficacy Study:

1. Age>=18, CHADS2 score>=1
2. Patients cannot be treated long-term with Warfarin
3. Eligible for clopidogrel and aspirin
4. Provide written informed consent and agree to comply with the required follow-ups

Exclusion Criteria:

- Exclusion criteria: Patients who did not participate in the LAmbreTM Safety and Efficacy Study or did not complete 1-year follow-up LAmbreTM Safety and Efficacy Study.

The exclusion criteria of LAmbreTM Safety and Efficacy Study:

1. Need to take Warfarin
2. Presence of rheumatic, degenerative or congenital valvular heart diseases
3. Early stage or paroxysmal atrial fibrillation
4. Symptomatic patients with carotid artery disease (such as carotid stenosis>=50%)
5. Heart failure NYHA grade IV
6. Recent 30 days stroke or TIA
7. Presence of active sepsis or endocarditis
8. Cardiac tumours or other malignancy with estimated life expectancy <2 years
9. Abnormal blood test; renal dysfunction
10. LAA removed or heart implant patients
11. Patients have planned electrophysiological ablation or cardioversion 30 days post implantation of the LAmbre system
12. Patients have a history of mechanical prosthesis operation
13. Patients who are pregnant, or desire to be pregnant during the during the study
14. Participation in other trials
15. A known allergy to nitinol
16. Patients will not be able to complete the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated in the LAmbreTM Safety and Efficacy Study and completed the 1-year follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2018-11-20 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of compound event | 5 years after the surgery
  The compound event including death, systemic embolization, complications related to the device and requiring treatment (cardiac embolism, embolization, stroke, hemorrhage, death).

SECONDARY OUTCOMES:
The incidence of MACCE events | 2,3,4,5 years postoperative follow-up.
  The MACCE events including death (All cause death, All-cause death includes cardiac death, non-cardiac death and unexplained death), stroke, cardiac tamponade, and renal failure.
Ischemic stroke rate | 2,3,4,5 years postoperative follow-up
  Ischemic stroke is a neurological deficit caused by transient ischemic attack, cerebral thrombosis or cerebral embolism.
The rate of stroke | 2,3,4,5 years postoperative follow-up
  Stroke is deviated into ischemic, hemorrhagic or undetermined stroke, and transient ischemic attacks (TIA).
The event of bleeding | 2,3,4,5 years postoperative follow-up
  Intracranial or alimentary canal, or any bleeding that requires transfusion of 2 units of red blood cell suspension.
Cardiac events | 2,3,4,5 years postoperative follow-up
  Non-fatal myocardial infarction, arrhythmia, cardiac tamponade, cardiogenic shock, endocarditis.

CONTACTS AND LOCATIONS:
Overall Officials: Congxin Huang, Principal Investigator — People's Hospital of Wuhan University
Locations (11):
- China (11):
  - Beijing Chaoyang Hospital, Capital Medical university, Beijing, Beijing Municipality
  - Fuwai Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Shandong
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu